CLINICAL TRIAL: NCT04918017
Title: Treatment Outcomes For Functional Dyspepsia Based On Current International Guidelines In Multi-Ethnic Asian Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Chuah Kee Huat, Principal Investigator, Clinical Specialist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345676
Record Dates: First submitted 2021-05-04; First posted 2021-06-08 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Functional Dyspepsia
Keywords: Itopride; Proton Pump Inhibitor; Functional dyspepsia; FGID
MeSH Terms: interventions — itopride; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment based on subtypes: Epigastric Pain Syndrome (EPS) (Experimental): EPS: treat with esomeprazole 40mg OD (proton pump inhibitor)
  Interventions: Drug: Treatment based on subtypes: Esomeprazole or Itopride
- Treatment based on subtypes: Post Prandial Distress Syndrome (PDS) (Experimental): PDS: treat with itopride 50mg TDS (prokinetic)
  Interventions: Drug: Treatment based on subtypes: Esomeprazole or Itopride
- Treatment based on subtypes: Overlapped EPS/ PDS (Experimental): Overlapped EPS/PDS: treat with itopride 50mg TDS first and add esomeprazole 40mg OD (if partially responded) or change to esomeprazole 40mg OD (if not responded)
  Interventions: Drug: Treatment based on subtypes: Esomeprazole or Itopride
- Treatment with Proton Pump Inhibitor regardless of subtype (Active Comparator): Treat with esomeprazole 40mg OD (proton pump inhibitor) regardless of subtype of functional dyspepsia
  Interventions: Drug: Treatment with proton pump inhibitor regardless of subtype: Esomeprazole

INTERVENTIONS:
Drug: Treatment based on subtypes: Esomeprazole or Itopride — Esomeprazole 40mg OD for EPS and Itopride 50mg TDS for PDS
  In overlapped EPS/ PDS: treat with Itopride 50mg TDS first and then add Esomeprazole 40mg OD (if partially responded- assessed at week 4) or treat with Itopride 50mg TDS first and then change to Esomeprazole 40mg OD (if not responded- assessed at week 4)
  Arms: Treatment based on subtypes: Epigastric Pain Syndrome (EPS); Treatment based on subtypes: Overlapped EPS/ PDS; Treatment based on subtypes: Post Prandial Distress Syndrome (PDS)
Drug: Treatment with proton pump inhibitor regardless of subtype: Esomeprazole — Esomeprazole 40mg OD
  Arms: Treatment with Proton Pump Inhibitor regardless of subtype

SUMMARY:
Functional dyspepsia (FD) is among the most established and common functional gastrointestinal disorders (FGIDs). FD is subdivided into two subtypes based on symptoms: epigastric pain syndrome (EPS) and postprandial distress syndrome (PDS).

Based on international guidelines (Asian Consensus and Rome Consensus), a prokinetic, medication which promotes gut movement (such as Itopride) should be the 1st line treatment for the PDS sub-type and a proton pump inhibitor, medication which reduces stomach acid production (such as Esomeprazole) should be the 1st line treatment for the EPS sub-type.

However, in the routine practice in Malaysia, proton pump inhibitor is still commonly used as 1st line treatment for FD, regardless of subtypes. This may be one of the reasons why FD continues to be inadequately treated locally and causes poor health-related quality of life (QOL) in FD patients.

The purpose of this study is to compare the clinical symptoms and quality of life improvement in patients with functional dyspepsia (FD) after treatment according to international guidelines versus treatment according to routine practice. Adverse effects when managed according to guidelines versus routine practice will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Functional Dyspepsia using Rome IV diagnostic criteria: patients on prior dyspepsia treatment can be recruited after washout period of 2 weeks
2. Subject who has ability to provide written informed consent and willingness to comply with the requirement of the protocol
3. Able to communicate in English, Malay or Mandarin languages

Exclusion Criteria:

1. Patients with known hypersensitivity to Itopride and/or proton pump inhibitors or to any of the excipients of the study medication
2. Patients with a contraindication to any of the study drugs
3. Pregnant / breast feeding women
4. Presence of family history of GI malignancy or alarm features suggested malignancy - e.g. Unintentional weight loss (≥ 10% of body weight in recent 6 months), GI bleeding
5. Patients consuming regular Aspirin or NSAIDs (except low-dose Aspirin at a dose of 325 mg/day or less for cardiovascular prophylaxis)
6. History of erosive esophagitis, peptic ulcer disease within 1 year prior to the screening
7. History of gastrointestinal (GI) malignancy, primary esophageal motility disorder, documented upper GI surgery
8. Patients with any hepatobiliary or pancreatic diseases
9. Patients with severe depression, anxiety, or other psychological disorder
10. Patients with any terminal disease
11. Presence of irritable bowel syndrome (Rome IV criteria) or inflammatory bowel disease (IBD)
12. Other conditions determined by the investigator to be inappropriate for this clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Global symptom change in patients with FD when managed according to guidelines, compare to routine practice | 8 weeks
  Assessment of global symptom change using 'Overall Treatment Effect' (OTE) questionnaire from baseline to 8 weeks of treatment.
  Patients who were 'extremely improved' or 'improved' on the OTE scale are considered responders. This will be compared with intervention arm and routine practice arm.

SECONDARY OUTCOMES:
Individual upper gastrointestinal (UGI) symptoms change | 8 weeks
  Change in individual upper gastrointestinal (UGI) symptoms (total 9 symptoms). Patients will be assessed on nine UGI symptoms (upper abdominal pain, upper abdominal discomfort, postprandial fullness, upper abdominal bloating, early satiety, excessive belching, nausea, vomiting and heartburn) and they will rate each symptom on a severity scale of 0-3 (none, mild, moderate and severe).
  On assessment of individual symptoms, patients who have a decrease in symptom severity of ≥50% from baseline are considered responders. Nine individual symptoms are evaluated and compared between intervention and routine practice group.
Change of quality of life | 8 weeks
  The change in Health-Related Quality of Life (HRQOL) score based on Short Form-Napean Dyspepsia Index Questionnaire (SF-NDI).
  It is a 10-item questionnaire with 5 sub-scales each examining the influence of dyspepsia on domains of health in patients, namely tension/anxiety, interference with daily activities, disruption to regular eating/drinking, knowledge towards/control over disease symptoms and interference with work/study, with each sub-scale containing two items [10]. Each item is measured by a 5-point Likert scale ranging from 0 (not at all or not applicable), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely). Individual items in each sub-scale are aggregated to obtain a score range from 0 (lowest HRQoL score) to 100 (highest HRQoL score) as per the developers' original calculation formula. A total, overall SF-NDI total score is obtained using the mean of 5 subscale scores.
Incidence of Adverse effects | 12 weeks
  Incidence of adverse events of treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Huat Chuah, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuah KH, Loo QY, Hian WX, Khoo XH, Panirsheeluam S, Jubri NBM, Natarajan V, Khoo S, Mahadeva S. Clinical Trial: Treatment of Functional Dyspepsia According to Subtype Compared With Empirical Proton Pump Inhibitor. Aliment Pharmacol Ther. 2025 Jan;61(2):258-267. doi: 10.1111/apt.18418. Epub 2024 Dec 2. PMID 39618195